CLINICAL TRIAL: NCT01676506
Title: The Impact of Genetic Polymorphisms on Ranibizumab Treatment Outcomes in Wet Age-Related Macular Degeneration (AMD)
Brief Title: Genetic Polymorphisms in Ranibizumab Treatment in Wet Age-Related Macular Degeneration (AMD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ekaterina Chikun, Researcher, Russian Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GB-1000-LC
Record Dates: First submitted 2012-01-17; First posted 2012-08-31 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Age-Related Macular Degeneration
Keywords: Wet AMD; genetic polymorphisms; Ranibizumab
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal injections of 0.5mg/0.05 mL dosage, injected at months 0, 1, and 2.
  Other Names: Lucentis
Procedure: Ranibizumab Injection

SUMMARY:
Genetic factors of an individual patient may have an impact on Ranibizumab (Lucentis) treatment outcome in patients with Wet Age-Related Macular Degeneration (AMD).

DETAILED DESCRIPTION:
Age-Related Macular Degeneration (AMD) is a disease that affects central part of the retina, called macula, and is associated with progressive central vision loss. Moreover, AMD is known to be a leading cause of blindness in developed countries. In wet form of AMD, new abnormal blood vessels start to grow from the choroid towards the retina that leads to leakage from these vessels and, in turn, to impaired retinal structure and rapid vision loss.

Genetic factors were found to be important in development of wet AMD. Our previous research showed the association between some genetic polymorphisms and the risk of wet AMD as well as with specific clinical features of the disease. At present, anti-vascular endothelial growth factor (anti-VEGF) therapy with intravitreous ranibizumab (Lucentis) is considered to be the most effective treatment for wet AMD. However, treatment outcomes may vary significantly from improved vision to no effect. The aim of this research is to study how ranibizumab treatment outcomes depend on genetic factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 50 years old
* Neovascular age-related macular degeneration
* CNV in the central part of the retina (macular is involved)
* Active CNM (seen on fundus fluorescein angiography)
* CNV activity is on one of the following: sub-retinal hemorrhage, sub-retinal lipid, documented loss of 3 lines of vision during last 3 months
* Visual acuity of between 20/40 and 20/300 (ETDRS)

Exclusion Criteria:

* Patients under 50 years old
* Patients with CNM not caused by AMD
* Patients physically unable to tolerate intravenous fluorescein angiography
* Patients with medically uncontrolled glaucoma
* Patients with history of bronchial asthma, thrombophlebitis, polyvalent allergy, cancer
* Any intraocular surgery within 3 months in the study eye
* Prior retinal or vitreous surgery including vitrectomy or scleral buckling
* Any significant ocular disease other than AMD that has compromised or could compromise vision in the study eye and confound analysis of the primary outcome
* Individuals with physical or mental disabilities that prevent accurate vision testing
* History of any laser treatment of CNV in study eye (laser photocoagulation or prior photodynamic therapy), or anti-VEGF (ranibizumab or bevacizumab) in the past 2 years in the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | Baseline and month 3
  Best corrected visual acuity will be assessed by standardized vision testing, early treatment diabetic retinopathy study (ETDRS) test.

CONTACTS AND LOCATIONS:
Overall Officials: Mariya Budzinskaya, MD, PhD, Study Chair — State Research Institute of Eye Disease of Russian Academy of Medical Sciences
Locations (1):
- State Research Institute of Eye Disease of Russian Academy of Medical Sciences, Moscow, Russia